CLINICAL TRIAL: NCT04822415
Title: Anaesthetic Efficacy of 2% Mepivacaine Versus 4% Articaine for Inferior Alveolar Nerve Blocks in Patients With Symptomatic Irreversible Pulpitis in Mandibular Molars: A Randomized Clinical Trial
Brief Title: Anaesthetic Efficacy of 2% Mepivacaine Versus 4% Articaine With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzan AW Amin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ENDO-CU-2014-06-09
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Mepivacaine; Carticaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mepivacaine (Experimental): IANB using 3.6 ml of 2% mepivacaine hydrochloride with 1:100,000 epinephrine.
  Interventions: Drug: Mepivacaine
- Articaine (Active Comparator): IANB using 3.4 ml of 4% articaine hydrochloride with 1:100,000 epinephrine.
  Interventions: Drug: Articaine

INTERVENTIONS:
Drug: Mepivacaine — IANB using 3.6 ml of 2% mepivacaine hydrochloride with 1:100,000 epinephrine.
  Arms: Mepivacaine
Drug: Articaine — IANB using 3.4 ml of 4% articaine hydrochloride with 1:100,000 epinephrine.
  Arms: Articaine

SUMMARY:
The aim of this randomized, double-blinded, clinical trial was to assess the effect of 3.6 mL 2% mepivacaine hydrochloride with 1:100,000 epinephrine compared to 3.4 mL 4% articaine hydrochloride with 1:100,000 epinephrine on the success of the inferior alveolar nerve block for patients with symptomatic irreversible pulpitis in mandibular molars.

DETAILED DESCRIPTION:
The aim of this randomized, double-blinded, clinical trial was to assess the effect of 3.6 mL 2% mepivacaine hydrochloride with 1:100,000 epinephrine compared to 3.4 mL 4% articaine hydrochloride with 1:100,000 epinephrine on the success of the inferior alveolar nerve block for patients with symptomatic irreversible pulpitis in mandibular molars. Patients were clinically and radiographically examined and their eligibility assessed and preoperative pain was measured using the numerical rating scale (NRS). Patients were randomly assigned to one of 2 groups: experimental group (2% mepivacaine) and the control group (4% articaine). After 15 minutes of the inferior alveolar nerve block (IANB), patients reporting lip numbness had their molars accessed. No-to-mild pain response was considered success during root canal preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health (American Society of Anesthesiologists Class I or II).
* Patients having symptomatic irreversible pulpitis in one of their mandibular molars.
* Age range between 18 to 50 years.
* Patients who can understand Numerical Rating Scale (NRS).
* Positive patient acceptance and the ability to sign an informed consent.

Exclusion Criteria:

* Pregnant females.
* Patients allergic to articaine, mepivacaine and/or any used medication or material.
* Patients having active sites of pathosis in the area of injection.
* Patients having active pain in more than one molar.
* Patients who had taken analgesics in the 12 hours preceding treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Anaesthetic success | Intraoperative
  Success of mandibular inferior alveolar nerve block anesthesia during access cavity preparation and instrumentation measured using the 11-point numerical rating scale (NRS) so that no-or-mild pain is considered as anesthetic success and moderate-to-severe pain is considered anesthetic failure.

SECONDARY OUTCOMES:
Need for Supplemental anaesthesia | Intraoperative
  The need for supplemental anaesthesia to complete treatment (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Randa ElBoghdadi, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allegretti CE, Sampaio RM, Horliana AC, Armonia PL, Rocha RG, Tortamano IP. Anesthetic Efficacy in Irreversible Pulpitis: A Randomized Clinical Trial. Braz Dent J. 2016 Jul-Aug;27(4):381-6. doi: 10.1590/0103-6440201600663. PMID 27652697
- [Background] Nagendrababu V, Pulikkotil SJ, Suresh A, Veettil SK, Bhatia S, Setzer FC. Efficacy of local anaesthetic solutions on the success of inferior alveolar nerve block in patients with irreversible pulpitis: a systematic review and network meta-analysis of randomized clinical trials. Int Endod J. 2019 Jun;52(6):779-789. doi: 10.1111/iej.13072. Epub 2019 Feb 12. PMID 30638269